CLINICAL TRIAL: NCT01458249
Title: An Open-label, Multicenter, Phase 2 Study to Evaluate the Efficacy and Safety of Eribulin Mesylate in Previously Treated Subjects With Advanced or Metastatic Soft Tissue Sarcoma
Brief Title: An Open-label, Multicenter, Phase 2 Study to Evaluate the Efficacy and Safety of Eribulin Mesylate in Previously Treated Subjects With Advanced or Metastatic Soft Tissue Sarcoma (Study E7389-J081-217)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7389-J081-217
Record Dates: First submitted 2011-10-21; First posted 2011-10-24 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Soft Tissue Sarcoma
Keywords: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — eribulin

ARMS (1):
- eribulin mesylate 1.4 mg/m^2 (Experimental)
  Interventions: Drug: eribulin mesylate

INTERVENTIONS:
Drug: eribulin mesylate — Administration of eribulin mesylate at a dose of 1.4 mg/m^2 as an IV bolus infusion over 2-5 minutes on Days 1 and 8 of every cycle, where the duration of each cycle is 21 days.
  Other Names: E7389

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of eribulin mesylate in subjects with soft tissue sarcoma who received at least one standard chemotherapy (an anthracycline or an ifosfamide monotherapy or a combination therapy).

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed soft tissue sarcoma of high or intermediate grade
* Documented evidence of advanced or metastatic soft tissue sarcoma, not amenable to surgery or radiotherapy
* Within 6 months from the radiographic evidence of disease progression by RECIST criteria in the last chemotherapy regimen for advanced or metastatic soft tissue sarcoma
* Presence of measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Subjects who received at least one standard chemotherapy for advanced soft tissue sarcoma (an anthracycline or an ifosfamide monotherapy, or a combination therapy)
* Subjects aged ≥ 20 years at the time of informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Adequate organ function
* Voluntary agreement to provide written informed consent

Exclusion Criteria

* A history of malignancies or recurrence within 5 years after the remission
* Significant cardiovascular impairment
* Any serious concomitant illness or infection requiring treatment.
* Hypersensitivity to either halichondrin B or halichondrin B chemical derivatives or both.
* Subjects who have previously participated in a study with eribulin (whether treated with eribulin or not).
* Any medical or other condition which, in the opinion of the principal investigator, will preclude participation in a clinical trial.
* Subjects who have received any anti-cancer therapy, including surgery, radiotherapy, immunotherapy, cytotoxic, hormonal, biological (including humanized antibodies) and targeted agents within 21 days, or any investigational agent within 30 days, prior to the first dose of study drug.
* Subjects who have not recovered from toxicities as a result of prior anti-cancer therapy to ≤ Grade 1, according to Common Terminology Criteria for Adverse Events (CTCAE), except for peripheral neuropathy of Grade 2 and alopecia.
* Subjects with known cerebral metastases with clinical symptoms or requiring treatment.
* Pre-existing peripheral neuropathy > CTCAE Grade 2.
* Female subjects must not be pregnant with a negative by the pregnancy test at Screening, or breastfeeding.
* Subjects participating in other clinical trials

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-11; Primary Completion 2014-11 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Obaishi, Study Director — Eisai Co., Ltd.
Locations (12):
- Japan (12):
  - Nagoya, Aichi-ken
  - Kashiwa, Chiba
  - Fukuoka, Fukuoka
  - Hidaka, Hokkaido
  - Sapporo, Hokkaido
  - Tsu, Mie-ken
  - Okayama, Okayama-ken
  - Osaka, Osaka
  - Suita, Osaka
  - Bunkyo, Tokyo
  - Chuo-ku, Tokyo
  - Shinjuku, Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- All Treated Participants (Arm 1 and Arm 2): Eribulin mesylate was administered at a dose of 1.4 mg/m^2 as an intravenous (IV) infusion over 2 to 5 minutes on Days 1 and 8 of every cycle, where the duration of each cycle is 21 days (3 weeks).
Period: Overall Study
Arm/Group | All Treated Participants (Arm 1 and Arm 2)
Started | 52
Participants Treated | 51
Completed | 44
Not Completed | 8
Not completed — Not treated | 1
Not completed — Adverse Event | 4
Not completed — Other | 2
Not completed — Ongoing | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who received at least one dose of study drug. Arm 1 included all participants with ADI or LMS. Arm 2 included all participants with OTH.
Groups:
- Arm 1: Participants With ADI or LMS: Eribulin mesylate was administered at a dose of 1.4 mg/m^2 as an intravenous (IV) infusion over 2 to 5 minutes on Days 1 and 8 of every cycle, where the duration of each cycle is 21 days (3 weeks). Adipocyte sarcoma (ADI) or Leiomyosarcoma (LMS)
- Arm 2: Participants With OTH: Eribulin mesylate was administered at a dose of 1.4 mg/m^2 as an intravenous (IV) infusion over 2 to 5 minutes on Days 1 and 8 of every cycle, where the duration of each cycle is 21 days (3 weeks). Other types of eligible soft tissue sarcoma (OTH)
- Total: Total of all reporting groups
Arm/Group | Arm 1: Participants With ADI or LMS | Arm 2: Participants With OTH | Total
Number analyzed (Participants) | 35 | 16 | 51
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.4 (12.11) | 50.4 (12.44) | 51.1 (12.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 6 | 28
  Male | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Rate at 12 Weeks (PFR12wks)
Description: The PFR at 12 weeks was the percentage of participants with progression-free survival (success) measured as a binary variable based on the tumor response assessed at Week 12 after the start of study treatment. Participants were considered a success if one radiological evaluation performed at least Week 12 after start of therapy indicated stable disease (SD), or complete response (CR) or partial response (PR), as defined according to Response Evaluation Criteria in Solid Tumor version 1.1 (RECIST v1.1); all other cases were considered as failures (including disease progression or death before the Week 12 evaluation, or had unknown disease status at Week 12). If new anticancer treatments were started before the Week 12 evaluation, participants were considered failures. A 2-sided 90% confidence interval (CI) was calculated using the exact method of binomial distribution.
Time Frame: Week 12
Population: Full analysis set included all participants who received at least one dose of study drug. This was the primary analysis set for all efficacy evaluations. Arm 1 included all participants with ADI or LMS. Arm 2 included all participants with soft tissue sarcomas other than ADI or LMS (OTH).
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: Participants With ADI or LMS | Arm 2: Participants With OTH
Number analyzed (Participants) | 35 | 16
Percentage of participants | 60.0 [44.7 to 74.0] | 31.3 [13.2 to 54.8]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival was defined as the time from the date of treatment start to the first documented date of event (disease progression or death from any cause, whichever occurred first). PFS was assessed every six weeks (until disease progression was confirmed, or sooner, if clinically indicated) and was based on Investigator and Independent Review Committee (IRC) assessments according to RECIST v1.1. Disease progression was measured using computed tomography (CT) or magnetic resonance imaging (MRI) on targeted tumors and defined as at least a 20% relative increase and 5 mm absolute increase in the sum of diameters of target lesions (taking as reference the smallest sum on study), recorded since the treatment started or the appearance of 1 or more new lesions. A 95% CI was calculated using Kaplan-Meier estimate and Greenwood Formula. A generalized Brookmeyer and Crowley method was used to construct a log-log-transformed 95% CI.
Time Frame: Cycle 1 (Day 1) to progressive disease (PD) or death, or date of study cutoff (14 Nov 2014) up to 3 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1: Participants With ADI or LMS | Arm 2: Participants With OTH
Number analyzed (Participants) | 35 | 16
Months | 5.52 [2.79 to 8.18] | 2.01 [1.22 to 4.07]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from the date of treatment start to the date of death from any cause. Participants were followed for survival every twelve weeks after PD. In the absence of confirmation of death, participants were censored either at the date that the participant was last known alive or the date of study cutoff, whichever came earlier. Participants censored before database cutoff included those who were lost to follow up and who withdrew consent. A 95% CI was calculated using Kaplan-Meier estimate and Greenwood Formula. A generalized Brookmeyer and Crowley method is used to construct a log-log-transformed 95% CI.
Time Frame: Cycle 1 (Day 1) to death, or date of study cutoff, (14 Nov 2014), up to 3 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1: Participants With ADI or LMS | Arm 2: Participants With OTH
Number analyzed (Participants) | 35 | 16
Months | 16.95 [11.01 to 20.47] | 7.64 [3.84 to 16.13]

4. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate was defined as the percentage of participants who had a best overall rate (BOR) of CR or PR. Tumor assessment was performed at Week 6 and Week 12 after the start of study treatment, and every six weeks thereafter. The BOR of CR and PR in this study required confirmation by a subsequent assessment of response at least four weeks (28 days) later. CR and PR were determined by the Investigator and IRC using RECIST v1.1 for target lesions assessed by MRI/CT scans. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had to have reduction in short axis to less than 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. A 95% CI was calculated using exact method of binomial distribution.
Time Frame: Date of CR or PR to the date of PD or death, whichever is first, or date of study cutoff (14 Nov 2014), up to 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: Participants With ADI or LMS | Arm 2: Participants With OTH
Number analyzed (Participants) | 35 | 16
Percentage of participants | 0 [0.0 to 10.0] | 0 [0.0 to 20.6]

5. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate was defined as the percentage of participants who had BOR of CR + PR + SD. BOR of SD must have manifested at least five weeks (35 days) after the first dose of study treatment. Tumor assessment was performed at Week 6 and Week 12 after the start of treatment, and every six weeks thereafter. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had to have reduction in short axis to less than 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of the longest diameter since the treatment started. A 95% CI was calculated using exact method of binomial distribution.
Time Frame: Date of CR, PR, or SD to date of PD or death, whichever is first, or date of study cutoff (14 Nov 2014), up to 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: Participants With ADI or LMS | Arm 2: Participants With OTH
Number analyzed (Participants) | 35 | 16
Percentage of participants | 80.0 [63.1 to 91.6] | 50.0 [24.7 to 75.3]

6. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR was defined as the percentage of participants who had a BOR of CR + PR + dSD (duration of SD greater than or equal to 11 weeks [77 days] after the first dose of study treatment). Tumor assessment was performed at Week 6 and Week 12 after the start of study treatment, and every six weeks thereafter. For participants whose BOR was SD, the duration of SD was defined as the time from the date of the first dose of study treatment to the first documented PD or death, whichever occurred first (i.e., same definition of PFS). If the dSD was censored at a time less than 11 weeks, the participant was considered as not having a clinical benefit. A 95% CI was calculated using exact method of binomial distribution.
Time Frame: First dose of study treatment to the date of CR, PR, or dSD to date of PD or death, whichever is first, or date of study cutoff (14 Nov 2014), up to 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: Participants With ADI or LMS | Arm 2: Participants With OTH
Number analyzed (Participants) | 35 | 16
Percentage of participants | 74.3 [56.7 to 87.5] | 50.0 [24.7 to 75.3]

7. Secondary Outcome: Durable Stable Disease (SD) Rate (dSDR)
Description: Durable stable disease rate was defined as the percentage of participants who manifested durable stable disease (the duration of stable disease for greater than or equal to eleven weeks) and was estimated based on the tumor response assessments performed according to RECIST v1.1. Tumor assessment was performed at Week 6 and Week 12 after the start of study treatment, and every six weeks thereafter. A 2-sided 95% CI was calculated using the exact method of binomial distribution.
Time Frame: Date of dSD to date of PD or death, whichever is first, or date of study cutoff (24 Nov 2014), up to 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: Participants With ADI or LMS | Arm 2: Participants With OTH
Number analyzed (Participants) | 35 | 16
Percentage of participants | 74.3 [56.7 to 87.5] | 50.0 [24.7 to 75.3]

8. Secondary Outcome: Best Overall Response (BOR)
Description: The best overall response categories (CR, PR, SD [including non-CR/non-PD], PD, not evaluable [NE], and unknown [UNK]) were derived based on time point tumor responses during the study as assessed by the IRC as well as the investigator. Tumor assessment was performed at Week 6 and Week 12 after the start of study treatment, and every six weeks thereafter. BOR of SD must have occurred at least 35 days (at least 5 weeks) after the first dose of study drug. If a participant had a BOR of non-CR/non-PD, the participant's BOR was grouped with the SD category.
Time Frame: Date of CR, PR, SD to PD or death of any cause, whichever is first, or date of study cutoff (14 Nov 2014), or up to 3 years
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: Participants With ADI or LMS | Arm 2: Participants With OTH
Number analyzed (Participants) | 35 | 16
Percentage of participants
  Complete response | 0 | 0
  Partial response | 0 | 0
  Stable disease | 80.0 | 50.0
  Progressive disease | 20.0 | 50.0
  Not evaluable | 0 | 0
  Unknown | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were collected beginning from the time of informed consent through 30 days after the last dose of study drug or until resolution, whichever came first. Participants were followed for an average of 18 weeks.
Description: Safety data was based on the safety analysis set which included all participants who received at least one dose of study drug and had at least one postbaseline safety evaluation. Treatment-emergent Serious AEs (SAEs) and non-serious AEs are reported in the safety section.
Arm/Group | All Treated Participants (Arm 1 and Arm 2)
Serious Adverse Events (participants affected / at risk) | 15/51
Other Adverse Events (participants affected / at risk) | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Treated Participants (Arm 1 and Arm 2) (N=51)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cataract (Eye disorders) | 1
Ileus (Gastrointestinal disorders) | 2
Hepatic haemorrhage (Hepatobiliary disorders) | 1
Infectious pleural effusion (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Streptococcal infection (Infections and infestations) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Tumour embolism (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Treated Participants (Arm 1 and Arm 2) (N=51)
Anaemia (Blood and lymphatic system disorders) | 24
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 51
Lymphopenia (Blood and lymphatic system disorders) | 40
Neutropenia (Blood and lymphatic system disorders) | 50
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Tachycardia (Cardiac disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 3
Cheilitis (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 16
Diarrhoea (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 21
Stomatitis (Gastrointestinal disorders) | 13
Vomiting (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 9
Malaise (General disorders) | 20
Oedema peripheral (General disorders) | 5
Pyrexia (General disorders) | 21
Hepatic function abnormal (Hepatobiliary disorders) | 5
Gingivitis (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 11
Upper respiratory tract infection (Infections and infestations) | 11
Urinary tract infection (Infections and infestations) | 3
Fall (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 14
Aspartate aminotransferase increased (Investigations) | 13
Blood alkaline phosphatase increased (Investigations) | 5
Blood creatine phosphokinase increased (Investigations) | 8
Blood lactate dehydrogenase increased (Investigations) | 11
C-reactive protein increased (Investigations) | 6
Weight decreased (Investigations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 12
Hyperlipidaemia (Metabolism and nutrition disorders) | 4
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10
Hypocalcaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 8
Hypoproteinaemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 7
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21
Dysgeusia (Nervous system disorders) | 12
Headache (Nervous system disorders) | 6
Neuropathy peripheral (Nervous system disorders) | 16
Peripheral sensory neuropathy (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 5
Proteinuria (Renal and urinary disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 14
Eczema (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 6
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other